CLINICAL TRIAL: NCT00878735
Title: The Effects of an Intensive Mindfulness Practice (Sesshin) on Neural Systems: an fMRI Evaluation of Healthy Volunteers and Cancer Patients
Brief Title: The Effects of a Meditation Retreat on Healthy Volunteers and Cancer Patients: an fMRI Study
Acronym: Sesshin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Elisa Kozasa, PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sesshin; Elisa
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Healthy; Cancer
Keywords: Meditation; Mindfulness; fMRI; cancer; stress; anxiety; depression; attention; Neuroscience; Neuroimaging; Psychobiology; Healthy volunteers (regular meditators and non-meditators)
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Zen meditation
  Interventions: Behavioral: Zen meditation
- 2 (No Intervention): No meditation (no intervention; keep regular activities) or a resting group (this group stays at the same place of the retreat group, but only to rest)

INTERVENTIONS:
Behavioral: Zen meditation — Zen meditation retreat (7 days: 5 days from 5:30 to 9:30 plus one day for adaptation and the departure day). The program starts everyday at 5:30 and finish at 9:30. In silence, the volunteers perform seating and walking meditation, stretching exercises, eating and all tasks in mindfulness.
  Other Names: Control group: no intervention
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the effects of a Zen meditation retreat (Sesshin) on psychophysiological parameters in healthy volunteers (regular meditators and non-meditators) and in cancer patients and to observe possible changes in the attentional circuitry (through functional Magnetic Resonance Imaging- fMRI) and in psychological tests (Beck Anxiety and Depression Inventories, Self-Compassion Scale, Mindfulness Attention Awareness Scale, Lipp Stress Scale for Adults).

DETAILED DESCRIPTION:
Meditation results in changes in cognition, sensory perception, affect, hormones, and autonomic activity. Until today, there have been very few imaging studies of the neural correlates of meditation. Instead of evaluating the meditation practice itself, our approach is to evaluate the neural correlates of performance modulation on an attention paradigm (the Stroop word-color task; SWCT) and an emotional paradigm (the frustration paradigm) before and after a meditation retreat. The following categories of individuals will be invited to participate: healthy regular meditation practitioners (at least three years of practice, three times a week), individuals inexperienced in meditation, and patients with a cancer diagnosis. The total sample will comprise 96 individuals who will be allocated to groups of sesshin meditation, rest groups and groups that will keep their daily activities. If they wish to do so, those who participate in the two latter groups may also receive training on meditation. The subjects will be between 18 and 65 years old and have no contraindication to the fMRI exam. After signing an informed consent form, the subjects will answer anxiety, depression and stress inventories; scales that evaluate their feelings of self-compassion and mindfulness, as well as the Stroop Color Word task and an emotional paradigm of functional Magnetic Resonance Imaging.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Men or women
* Left-handed or right-handed, as long as there are left-handed individuals in both groups for comparison
* Ages between 18 and 65
* No history of neurological or psychiatric problems, or use of controlled medication that might interfere with attention
* No symptoms of claustrophobia
* Written informed consent form to participate in the study

Cancer patients:

* The same criteria that apply to healthy volunteers in addition to a diagnosis of neoplasia confirmed by biopsy
* Volunteers should be undergoing post-therapeutical control, have no cure criteria yet, and not have been submitted to radio- or chemotherapy in the last three months

Exclusion Criteria:

Healthy Volunteers:

* Chemical dependence, including nicotine and alcohol
* Dementia or psychotic condition (established by a questionnaire)
* Depression or use of antidepressants
* Non-controlled severe organic disease that might interfere with the performance of the study, such as neoplasias, cardiopathies, digestive pathologies, diabetes mellitus type I or type II
* Neoplasias in the central nervous system
* Tremor or dystonia in cephalic segment that hinders the performance of the RMf study (tremor equal to or higher than 3 in each corporal segment, according to the UPDRS scale)
* Fulfillment of any criterion of contraindication for the MR exam (for instance, use of pacemaker; intracranial aneurism clip; cochlear implants)
* Presence of odontological devices that might disturb the magnetic field or any sources of variation of the magnetic susceptibility
* Presence of lesion in the encephalic parenchyma in the structural images. Exception is made to discreet punctiform areas in the white matter or a discreet reduction in the encephalic volume.
* Any other conditions the investigator might deem problematic for the inclusion of the volunteer in a trial of this nature will also be considered

Cancer patients:

* All the healthy volunteers, except for those that fit in the item: "non-controlled severe organic disease that might interfere in the performance of the study, such"
* The use of medication that acts on the central nervous system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the neural correlates of performance modulation on an attention paradigm (the Stroop word-color task; SWCT) and on an emotional paradigm (the frustration paradigm) before and after a Zen meditation retreat. | 2 years

SECONDARY OUTCOMES:
Anxiety, stress and depression symptoms, self-compassion feelings and mindfulness state will also be evaluated in healthy volunteers and cancer patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elisa H Kozasa, PhD, Principal Investigator — Instituto Israelita de Ensino e Pesquisa Albert Einstein
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Kozasa EH, Radvany J, Barreiros MA, Leite JR, Amaro E Jr. Preliminary functional magnetic resonance imaging Stroop task results before and after a Zen meditation retreat. Psychiatry Clin Neurosci. 2008 Jun;62(3):366. doi: 10.1111/j.1440-1819.2008.01809.x. No abstract available. PMID 18588603
- [Result] Kozasa EH, Sato JR, Lacerda SS, Barreiros MA, Radvany J, Russell TA, Sanches LG, Mello LE, Amaro E Jr. Meditation training increases brain efficiency in an attention task. Neuroimage. 2012 Jan 2;59(1):745-9. doi: 10.1016/j.neuroimage.2011.06.088. Epub 2011 Jul 7. PMID 21763432